CLINICAL TRIAL: NCT01604928
Title: A Randomized, Double-blind, Parallel Group, Proof of Concept Study of YM178 in Comparison With Placebo and Tolterodine in Patients With Symptomatic Overactive Bladder
Brief Title: Study to Test the Efficacy and Safety of YM178 in Subjects With Symptoms of Overactive Bladder
Acronym: Blossom
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 178-CL-008
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Urinary Bladder, Overactive
Keywords: Overactive Bladder; YM178; Mirabegron; Frequency; Urinary urge incontinence; Urgency; Urinary incontinence; Micturition
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Incontinence | interventions — mirabegron; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- YM178 Dose 1 (Experimental): low dose
  Interventions: Drug: YM178
- YM178 Dose 2 (Experimental): high dose
  Interventions: Drug: YM178
- Tolterodine (Active Comparator): Oral
  Interventions: Drug: tolterodine
- Placebo (Placebo Comparator): Oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YM178 — Oral
  Other Names: mirabegron
  Arms: YM178 Dose 1; YM178 Dose 2
Drug: tolterodine — Oral
  Other Names: Detrusitol
  Arms: Tolterodine
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
The study is intended to test efficacy, safety and tolerability of two doses of YM178 against placebo and tolterodine to treat patients with symptoms of over active bladder.

DETAILED DESCRIPTION:
This is a multinational, multicenter, double-blind, double-dummy,

randomized, parallel group, placebo and active controlled phase II proof-of concept study. Patients are enrolled into a single-blind, 2-week placebo run in

period after which they are randomized to 4 weeks of double-blind

treatment with YM178 (low dose and high dose), placebo or tolterodine. Subsequently patients will be followed for an additional 2 weeks

with single-blind placebo treatment. There are 6 visits in total: visit 1 at

enrolment, visit 2 (baseline) after the 2-week placebo run-in, visits 3, 4 and 5

after 1, 2 and 4 weeks of double-blind treatment respectively, and visit 6

after a 2-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to complete the micturition diary correctly.
* Symptoms of overactive bladder (urinary frequency and urgency with or without incontinence) for ≥ 3 months

At randomization:

* Patient must experience frequency of micturition on average ≥ 8 times per 24-hour period during the 3-day micturition diary period
* Patient must experience at least 3 episodes of urgency (grade 3 or 4) with or without incontinence, during the 3-day micturition diary period

Exclusion Criteria:

* Pregnant women or women who intend to become pregnant during the study or women of childbearing potential who are sexually active and practicing an unreliable method of birth control or will be lactating during the study. Reliable contraceptive methods are intra-uterine devices, contraceptive pills of combination type, hormonal implants, contraceptive patches and injectable contraceptives
* Clinically significant outflow obstruction (at the discretion of the investigator)
* Significant post void residual volume (PVR>200ml)
* Significant stress incontinence or mixed stress/urge incontinence where stress is the predominant factor as determined by the investigator (for female patients confirmed by a cough provocation test)
* Patients with a neurological cause for abnormal detrusor activity
* Diabetic neuropathy
* Evidence of a symptomatic urinary tract infection, chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy or previous or current malignant disease of the pelvic organs
* Uncontrolled narrow angle glaucoma, urinary or gastric retention, colitis ulcerosa, toxic megacolon, myasthenia gravis or any other medical condition which in the opinion of the investigator makes the use of anticholinergics contra-indicated
* Non-drug treatment including electrostimulation therapy

(a bladder training program or pelvic floor exercises which started more than 1 month prior to entry into the study can be continued)

* Use of medications intended to treat urinary incontinence or listed in Appendix 1 Part A. Part B lists medications that are restricted but accepted under certain conditions
* Known or suspected hypersensitivity to tolterodine, other anticholinergics, ß-adrenoceptor agonists, or lactose or any of the other inactive ingredients
* Any clinically significant cardiovascular complication including CVA, recent myocardial infarction and uncontrolled hypertension, indicated by a sitting systolic blood pressure ≥ 180 mmHg and/or diastolic blood pressure ≥ 110 mmHg
* Any clinically significant condition, which in the opinion of the investigator makes the patient unsuitable for the trial
* Participation in any clinical trial within 30 (90 in the UK) days prior to randomization
* Employees of the sponsor, third parties associated with the study, or the study site

At randomization:

* Patient who did not complete the micturition diary according to the instructions
* Average total daily urine volume > 3000 ml as recorded in the micturition diary
* Clinically significant elevation of serum creatinine or liver enzymes as evidenced by creatinine >150 mmol/L, ASAT or ALAT > 2x upper limit of normal range (ULN), γ-GT > 3x ULN and/or abnormal serum total bilirubin (as assessed in visit 1 samples or alternative sampling within 4 weeks prior to visit 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2004-04-05 (Actual); Primary Completion 2005-01-25 (Actual); Study Completion 2005-01-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean number of micturitions per 24 hours | Baseline and 4 weeks (end of treatment)

SECONDARY OUTCOMES:
Change from baseline in mean number of urgency episodes/24 hours | Baseline and 4 weeks (end of treatment)
Change from baseline in mean volume voided per micturition | Baseline and 4 weeks (end of treatment)
Change from baseline in mean number of urge incontinence episodes/24 hours | Baseline and 4 weeks (end of treatment)
Change from baseline in mean number of incontinence episodes/24 hours | Baseline and 4 weeks (end of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Director — Astellas Pharma Europe B.V.
Locations (30):
- Belgium (4):
  - Site: 12, Brussels
  - Site: 13, Edegem
  - Site: 11, Ghent
  - Site: 10, Leuven
- Czechia (6):
  - Site: 25, Mělník
  - Site: 22, Prague
  - Site: 24, Prague
  - Site: 20, Prague
  - Site: 21, Ústí nad Labem
  - Site: 23, Ústí nad Labem
- Germany (7):
  - Site: 32, Bad Ems
  - Site: 30, Emmendingen
  - Site: 35, Frankfurt
  - Site: 34, Hagenow
  - Site: 33, Hamburg
  - Site: 36, Koblenz
  - Site: 31, Trier
- Spain (3):
  - Site: 42, Alzira-Valencia
  - Site: 40, Madrid
  - Site: 43, Miranda de Ebro
- Sweden (5):
  - Site: 55, Gothenburg
  - Site: 53, Linköping
  - Site: 50, Lund
  - Site: 51, Stockholm
  - Site: 52, Uppsala
- United Kingdom (5):
  - Site: 64, Bimingham
  - Site: 62, London
  - Site: 63, London
  - Site: 60, Sheffield
  - Site: 61, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Chapple CR, Amarenco G, Lopez Aramburu MA, Everaert K, Liehne J, Lucas M, Vik V, Ridder A, Snijder R, Yamaguchi O; BLOSSOM Investigator Group. A proof-of-concept study: mirabegron, a new therapy for overactive bladder. Neurourol Urodyn. 2013 Nov;32(8):1116-22. doi: 10.1002/nau.22373. Epub 2013 Feb 19. PMID 23424164
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=194